CLINICAL TRIAL: NCT02806583
Title: Talking Time: Telephone Support Groups for Informal Caregivers of People With Dementia: A Randomized Controlled Trial
Brief Title: Talking Time: Telephone Support Groups for Informal Caregivers of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leipzig (Other)
Collaborators: German Center for Neurodegenerative Diseases (DZNE) (Other)
Responsible Party: Principal Investigator, Dr. Martin Berwig, Project Leader, University of Leipzig
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 932 000 - 151
Record Dates: First submitted 2016-06-09; First posted 2016-06-20 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Caregivers of People With Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): telephone based structured support groups
  Interventions: Other: structured support groups
- control (No Intervention): Active Comparator: Usual care (intervention as experimental group after 3 month (after T1)

INTERVENTIONS:
Other: structured support groups — Telephone-based Support Groups, information booklet and telephone-based preparatory meeting prior to the telephone-based support groups
  Arms: intervention

SUMMARY:
Caring for people with dementia (PwD) at home requires an enormous amount of time, organization and commitment. Therefore, informal caregivers (ICs), mainly relatives, of PwD often feel a high burden. Even though support groups on-site have shown positive effects on the subjective well-being and on the perceived social support of ICs, relatives either have no time or opportunity to leave the PwD alone or there are no support groups in the vicinity. The Talking Time project therefore aims to close this supply gap by providing structured telephone-based support groups in Germany for the first time. International studies have shown resulting benefits for ICs.

Methods/Design: The project will be evaluated in a cluster adjusted randomized controlled trial. The effects of the 3-months Talking Time intervention will be compared to a normal care group. Outcomes will be measured at two different times (baseline = T0, after 3 months =T1). The control group will receive the Talking Time intervention after T1.

ICs are eligible if they are 18 or older, have cared for the PwD for at least four hours on four days per week in the last six months. Exclusion criteria are psychiatric disorders of the IC.

Primary outcome of the effectiveness elevation is the subjective well-being of the relatives measured by the mental component of the SF-12. Secondary outcomes are the physical component summary of the SF-12, the Perceived Social Support Caregiver Scale, the Caregiver Reaction Scale and the Neuropsychiatric Inventory. For the process evaluation different quantitative and qualitative data sources will be collected addressing reach, fidelity, and dosage.

ELIGIBILITY:
Inclusion Criteria:

* medical ICD-10 dementia diagnosis available for the patient (F00.-*: Alzheimer disease or related disorders, F01.-: Vascular dementia, F03.-:Unspecified dementia)
* living with or sharing cooking facilities with the care recipient or providing care for a relative with diagnosed Alzheimer disease or related disorders for at least 4 hours on at least 4 days of a week for at least the past 6 months, respectively
* access to a telephone connection to be able to participate in the talking Time Intervention and the telephone- based interviews for the evaluation

Exclusion Criteria:

* lack of knowledge of German Language of informal caregiver
* risk of suicide in the informal caregiver
* actual psychiatric diagnosis of mental illness of the caregiver
* ICD-10-diagnosis of Dementia in other diseases classified elsewhere (F02.-*), except Dementia in Primary Parkinson disease (F02.3*) and Lewy Body disease (F02.8/G31.82)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11; Primary Completion 2017-03-13 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Mental Component Summary of the General Health Questionaires Short Form 12 (SF-12) | 3 months
  psychological quality of life of the caregivers

SECONDARY OUTCOMES:
Physical Component Summary of the SF-12 | 3 months
  physical quality of life of the caregivers
Perceived Social Support Caregiving Scale | 3 months
  perceived social Support of the caregivers
Caregiver Reaction Scale | 3 months
  caregivers burden
Neuropsychiatric Inventory | 3 months
  neuropsychiatric symptoms of patients

OTHER OUTCOMES:
General Practitioner assessment of COGnition (GPCOG) | Baseline
  cognitive abilities of Patient - Proxy rating
Functional Activities Questionnaire | 3 months
  functional activities ability of patients
  functional activities ability of patients - proxy rating
Patient Health Questionaire - 9 items (PHQ-9) | Baseline
  depression of caregivers

CONTACTS AND LOCATIONS:
Overall Officials: Martin Berwig, Dr., Principal Investigator — University of Leipzig
Locations (1):
- University of Leipzig, Leipzig, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Fraile E, Ballesteros J, Rueda JR, Santos-Zorrozua B, Sola I, McCleery J. Remotely delivered information, training and support for informal caregivers of people with dementia. Cochrane Database Syst Rev. 2021 Jan 4;1(1):CD006440. doi: 10.1002/14651858.CD006440.pub3. PMID 33417236
- [Derived] Dichter MN, Albers B, Trutschel D, Strobel AM, Seismann-Petersen S, Wermke K, Halek M, Berwig M. TALKING TIME: A pilot randomized controlled trial investigating social support for informal caregivers via the telephone. BMC Health Serv Res. 2020 Aug 25;20(1):788. doi: 10.1186/s12913-020-05523-9. PMID 32838773
- [Derived] Berwig M, Dichter MN, Albers B, Wermke K, Trutschel D, Seismann-Petersen S, Halek M. Feasibility and effectiveness of a telephone-based social support intervention for informal caregivers of people with dementia: Study protocol of the TALKING TIME project. BMC Health Serv Res. 2017 Apr 17;17(1):280. doi: 10.1186/s12913-017-2231-2. PMID 28415999